CLINICAL TRIAL: NCT05910567
Title: A Randomized Controlled Trial of Abdominal Ultrasound (FAST) in Children With Blunt Torso Trauma
Brief Title: A Research Study of Abdominal Ultrasound (FAST) in Children With Blunt Torso Trauma
Acronym: FAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Pediatric Emergency Care Applied Research Network (Network); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1943798; R01HD102571 (NIH)
Record Dates: First submitted 2023-05-09; First posted 2023-06-18 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Blunt Trauma to Abdomen; Wounds and Injuries; Abdomen Injury; Abdominal Injury; Abdomen, Acute
Keywords: Child; Wounds and Injuries; Blunt Trauma to Abdomen; Abdomen Injury; Blunt Abdominal Trauma
MeSH Terms: conditions — Wounds and Injuries; Abdominal Injuries; Abdomen, Acute | interventions — Ultrasonography; Physical Examination

STUDY DESIGN:
Intervention Model Description: Patients meeting enrollment criteria will be randomized to the FAST examination arm or to a standard of care/non-FAST examination arm using computer randomized order of enrollment. Randomization will be stratified by site and age group. Age groups will consist of participants 0 to their 3rd birthday and participants 3 years of age up to their 18th birthday. A minimum of 794 participants will be enrolled in the 0 to younger than 3 years of age group. To ensure concealment, opaque envelopes will be prepared at each study site using the randomization scheme provided by the lead institution. These envelopes will be readily available in the ED, provide the investigator with the randomized assignment, and contain the appropriate data collection form.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focused Assessment with Sonography for Trauma (FAST) Examination Arm (Other): Patients in this arm will under the FAST examination (abdominal ultrasound) for diagnostic purposes to detect the presence of blood in injured patients with blunt abdominal trauma.
  Interventions: Diagnostic Test: Focused Assessment with Sonography for Trauma (FAST) Examination
- No Intervention - Standard of Care - Without the FAST Examination (Other): Institution will use their standard operating procedures to deliver the usual care for injured patients with blunt abdominal/torso trauma.
  Interventions: Other: No Intervention: Standard of Care - Without the FAST Examination

INTERVENTIONS:
Diagnostic Test: Focused Assessment with Sonography for Trauma (FAST) Examination — A bedside Focused Assessment with Sonography for Trauma (FAST) Examination will be conducted on those participants who are randomized to the FAST arm.
  Other Names: Abdominal Ultrasound
  Arms: Focused Assessment with Sonography for Trauma (FAST) Examination Arm
Other: No Intervention: Standard of Care - Without the FAST Examination — Participants randomized to usual care will be evaluated per the standard operating procedures of the institution/site for the condition under study without the FAST exam.
  Arms: No Intervention - Standard of Care - Without the FAST Examination

SUMMARY:
Bleeding from intra-abdominal injuries is a leading cause of traumatic deaths in children. Abdominal CT is the reference standard test for diagnosing intra-abdominal injuries. Compelling reasons exist, however, to both aggressively evaluate injured children for intra-abdominal injuries with CT and to limit abdominal CT evaluation to solely those at non-negligible risk. The focused assessment sonography for trauma (FAST) examination can help focus patient evaluation in just this manner by potentially safely decreasing abdominal CT use in low risk children. This research study is a multicenter, randomized, controlled trial to determine whether use of the FAST examination, a bedside abdominal ultrasound, impacts care in 3,194 hemodynamically stable children with blunt abdominal trauma. The overall objectives of this proposal are 1) to determine the efficacy of using the FAST examination during the initial evaluation of children with blunt abdominal trauma, and 2) to identify factors associated with abdominal CT use in children considered very low risk for IAI after a negative FAST examination. The long-term objective of the research is to determine appropriate evaluation strategies to optimize the care of injured children, leading to improved quality of care and a reduction in morbidity and mortality.

DETAILED DESCRIPTION:
Trauma is a leading cause of death in children in the US. Abdominal trauma accounts for 30% of all pediatric traumatic deaths, second only to traumatic brain injury. Although CT is the reference standard for diagnosing intra-abdominal injury, it is associated with ionizing radiation, inducing malignancies at an estimated rate of 1 per 500 abdominal CT scans in children <5 years and 1 per 600 scans in adolescents. Thus, CT use should be limited to those at non-negligible risk of intra-abdominal injury.

The Focused Assessment with Sonography for Trauma (FAST) examination has also evolved as a diagnostic test for the evaluation for intra-abdominal injury; however, it is used primarily in adults. The FAST examination uses abdominal ultrasonography to detect the presence of intraperitoneal fluid in injured patients. If intraperitoneal fluid is identified following a traumatic injury, this fluid is presumed to be blood (hemoperitoneum). The FAST examination for detection of hemoperitoneum in trauma consists of several images. These include a right hepatorenal interface (Morison's pouch), perisplenic view, and longitudinal and transverse views of the pelvis.

Potential advantages of initial ED evaluation of the injured child using the FAST examination include: 1) bedside evaluation during initial patient ED evaluation and resuscitation; 2) rapid completion of the diagnostic test (within 3-5 minutes); 3) performance of the test and interpretation of results by ED physicians or trauma surgeons caring for the child; 4) no radiation exposure; and 5) reduced patient-care costs compared to routine use of abdominal CT. In adults, a positive FAST examination is the best predictor of intra-abdominal injury. In two adult randomized controlled trials, the use of FAST demonstrated improved patient care by decreasing abdominal CT use, complications and costs. Although the sensitivity of the FAST exam for intra-abdominal injury is lower than CT, as a screening test, it may decrease the need for abdominal CT in both low risk injured adults and children.

The long-term objective of this research study is to determine appropriate evaluation strategies to optimize the care of injured children, leading to improved quality of care and a reduction in morbidity and mortality. The specific aims of this proposal are to: 1) perform a randomized, controlled trial of the FAST examination in injured children and compare the frequency of abdominal CT scanning between children who are randomized to the FAST and non-FAST arms; 2) identify if an evaluation strategy including the FAST examination results in a similar frequency of missed or delayed diagnoses of intra-abdominal injuries than a strategy without the FAST examination; and 3) identify patient, physician, and system factors associated with obtaining abdominal CT scans in patients considered low risk for intra-abdominal injuries by the clinician after a negative FAST examination. Such a study has the potential for significant impact in improving the lives of injured children, if found to be successful.

This randomized controlled trial will follow the methods of the one prior randomized controlled trial of FAST in injured children which enrolled 925 injured children at a single center. This study incorporate a total of six centers to increase the sample size and generalizability of the results.

ELIGIBILITY:
Children younger than 18 years of age (0 to 17.9999 years) with blunt abdominal trauma presenting to the participating EDs within 24 hours of the traumatic event will be eligible if the do not meet any exclusion criteria and meet any one of the following inclusion criteria.

Inclusion Criteria:

1. Blunt torso trauma resulting from a significant mechanism of injury:

   * Motor vehicle collision: greater than 60 mph, ejection, or rollover
   * Automobile versus pedestrian/bicycle: automobile speed > 25 mph
   * Falls greater than 20 feet in height
   * Crush injury to the torso
   * Physical assault involving the abdomen
2. Decreased level of consciousness (Glasgow Coma Scale (GCS) score 9-14 or below age-appropriate behavior) in association with blunt torso trauma
3. Blunt traumatic event with any of the following (regardless of the mechanism):

   * Extremity paralysis
   * Multiple long bone fractures (e.g., tibia and humerus fracture)
4. History and physical examination suggestive of blunt torso trauma of any mechanism (including mechanisms of injury of less severity than mentioned above)

Exclusion Criteria:

The following patients will be excluded from the study:

1. Age-adjusted low blood pressure (Hemodynamic instability)

   * Patients will be excluded for prehospital or initial age-adjusted ED low blood pressure. This is because the standard evaluation of these patients involves immediate FAST based on prior work by our group. Low blood pressure is determined based upon the patient's age, and will be defined as a systolic blood pressure less than 70 mm Hg for patients younger than 1 month, less than 80 mm Hg for ages 1 month to 5 years, and less than 90 mm Hg for ages over 5 years.
2. Penetrating trauma: Patients who are victims of stab or gunshot wounds
3. Traumatic injury occurring > 24 hours prior to the time of presentation to the ED
4. Transfer of the patient to the ED from an outside facility with abdominal CT scan, diagnostic peritoneal lavage, or laparotomy previously performed
5. Transferred with FAST exam already performed at outside hospital
6. Patients with known disease processes resulting in intraperitoneal fluid including liver failure and the presence of ventriculoperitoneal shunts
7. Initial GCS score ≤ 8 as it is standard for children with GCS scores ≤ 8 to undergo abdominal CT if blunt abdominal trauma is suspected
8. Known pregnancy
9. Known prisoner
10. Known intra-abdominal injury diagnosed within 30 days prior of this ED visit

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4346 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of abdominal CT scanning | For the duration of the subject's Emergency Department stay and initial hospitalization (up to 24 hours)
  The primary outcome is the rate of abdominal CT scanning in each study arm, measured for each patient categorically (yes/no) during the Emergency Department stay and initial hospitalization (up to 24 hours).
Rate of delayed or missed or delayed intra-abdominal injuries | In hospitalized participants, IAI collection will be captured from the time of assignment until discharge (up to 30 days). For participants discharged from the ED IAI collection will be captured from the time of assignment until 7 days after ED discharge
  The rate of missed or delayed intra-abdominal injuries (IAI) will be identified and reported for any cases with a delay in diagnosis (i.e., patients diagnosed with IAI in the hospital after ED disposition) or missed IAI (IAI diagnosed after discharge from the ED/hospital).
Identifying variables associated with obtaining abdominal CT scans in very low risk patients with normal FAST examinations | The binary indicator assessment of yes/no will occur upon discharge from the Emergency Department or admission to the hospital, an average of 6.5 hours
  This primary outcome will be a binary indicator (yes/no) for whether the patient with a normal FAST examination who is thought by the clinician to have less than a 1% risk of intra-abdominal injury nonetheless undergoes abdominal CT (outcome of interest).

SECONDARY OUTCOMES:
Emergency Department (ED) length of stay | ED length of stay will be calculated in minutes from the time of ED arrival until the time of ED discharge or the time from ED arrival until the time of hospital admission assessed up to 7 days.
  ED length of stay is a continuous variable measured in minutes. The investigators will compare the ED length of stay between study arms using nonparametric methods (time from ED arrival to hospital admission or time from ED arrival until ED discharge).
Rate of Hospitalization | The assessment of the categorical variable yes/no will occur upon the participants discharge from the Emergency Department or admission to the hospital, an average of 6.5 hours
  Rate of hospitalization is a categorical variable (yes/no) on whether the patient is hospitalized on initial, enrolling ED visit. The investigators will compare the rate of hospitalization between study arms using categorical statistical methods.
Physician suspicion of intra-abdominal injury | All physician suspicion assessments will occur up to 24 hours after a participants ED presentation
  Physician suspicion of intra-abdominal injury is collected after initial physician evaluation for all patients. For those patients who are randomized to the FAST examination this information is collected again after completing the FAST examination. Physician suspicion is collected as follows: Less than 1%, 1-5%, 6-10%, 11-50%, greater than 50%.
Rate of abdominal CT scanning in children 0 to 3 years of age. | For the duration of the subject's Emergency Department stay and initial hospitalization (up to 24 hours).
  In this prespecified age group, the outcome is the rate of abdominal CT scanning in each study arm, measured for each patient categorically (yes/no) during the Emergency Department stay and initial hospitalization (up to 24 hours).
Laparotomy (surgery to the abdomen) rate | For the first seven days after the time of injury.
  Laparotomy rate is a binary indicator (yes/no) for whether the patient underwent a laparotomy (surgery to the abdomen) to identify/repair an intra-abdominal injury.

CONTACTS AND LOCATIONS:
Overall Officials: James F Holmes, MD, MPH, Principal Investigator — University of California, Davis; Nathan Kuppermann, MD, MPH, Principal Investigator — University of California, Davis
Locations (6):
- United States (6):
  - University of California, Davis Medical Center, Sacramento, California
  - University of Colorado, Anschutz Medical Center and Children's Hospital Colorado, Aurora, Colorado
  - Emory University Children's Healthcare of Atlanta, Atlanta, Georgia
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holmes JF, Tancredi DJ, Kelley KM, Griffiths M, Gold DL, Lam SHF, Stone B, Brenkert T, Andrade AN, Hanson E, Gwal K, Kornblith A, Hirose S, Utter GH, Kuppermann N. Abdominal ultrasound (FAST) in hemodynamically stable children with blunt abdominal trauma: study protocol for a randomized controlled trial. Trials. 2025 Dec 12;26(1):564. doi: 10.1186/s13063-025-09137-6. PMID 41388553
- See also: Pediatric Emergency Care Applied Research Network — https://pecarn.org